CLINICAL TRIAL: NCT04428905
Title: Self-Management to Optimize Survivorship Care and Outcomes in Lung and Colorectal Cancers
Brief Title: Self-Management Survivorship Care in Stage I-III Non-small Cell Lung Cancer or Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19556; NCI-2020-03375 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19556 (Other: City of Hope Medical Center); R01CA249501 (NIH)
Record Dates: First submitted 2020-05-26; First posted 2020-06-11 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage I Colorectal Cancer AJCC v8; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Colorectal Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Colorectal Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage IIC Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Lung Neoplasms | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (personalized care plan, telehealth sessions) (Experimental): Patients receive a personalized care plan/resource manual. Patients also participate in 5 telehealth sessions with a nurse over 60 minutes each for 4 months (months 1-4) about self-management skills building, then 3 maintenance telehealth sessions with a nurse over 60 minutes each for 3 months (months 5-7) for additional self-management skills building support. A copy of patient's care plan is also sent to their PCP.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survivorship Care Plan; Other: Telemedicine
- Arm II (ASCO care plan, telehealth sessions) (Active Comparator): Patients receive an ASCO care plan. Patients also participate in 5 telehealth sessions with a nurse over 60 minutes each for 4 months (months 1-4) to answer questions on a handbook about life after cancer treatment, then 3 monthly telehealth sessions with a nurse over 60 minutes each for 3 months (months 5-7) to answer questions about the handbook. A copy of the ASCO care plan is also sent to their PCP.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Telemedicine

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Survivorship Care Plan — Receive personalized care plan/resource manual
  Arms: Arm I (personalized care plan, telehealth sessions)
Other: Telemedicine — Participate in telehealth sessions
  Other Names: Telehealth

SUMMARY:
This phase III trial studies how well a telehealth self-management program works in improving survivorship care and outcomes in stage I-III non-small cell lung cancer or colorectal cancer survivors. Survivor self-management program focuses on coaching patients on follow-up care after cancer treatments. Participating in the program may improve knowledge and confidence about follow-up care, communication with cancer care and primary care doctors, and quality of life after cancer treatment in non-small cell lung cancer or colorectal cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of the intervention on care coordination, communication, and primary care provider (PCP) knowledge, comparing the intervention and attention control arms at 4 and 8 months post-accrual.

II. Determine the efficacy of the intervention on survivor outcomes, comparing the intervention and attention control arms at 4 and 8 months post-accrual.

EXPLORATORY OBJECTIVE:

I. Assess the reach, efficacy, adoption, implementation, and maintenance (RE-AIM) of the intervention.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (SURVIVOR SELF-MANAGEMENT): Patients receive a personalized care plan/resource manual. Patients also participate in 5 telehealth sessions with a nurse over 60 minutes each for 4 months (months 1-4) about self-management skills building, then 3 maintenance telehealth sessions with a nurse over 60 minutes each for 3 months (months 5-7) for additional self-management skills building support. A copy of patient's care plan is also sent to their PCP.

ARM II (ATTENTION CONTROL): Patients receive an American Society of Clinical Oncology (ASCO) care plan. Patients also participate in 5 telehealth sessions with a nurse over 60 minutes each for 4 months (months 1-4) to review a handbook about life after cancer treatment, then 3 monthly telehealth sessions with a nurse over 60 minutes each for 3 months (months 5-7) to answer questions about the handbook. A copy of the ASCO care plan is also sent to their PCP. After study initiation, patients are followed up at 4 and 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer (NSCLC) and colorectal cancer survivors who are 4 months post-treatment completion
* History of stage I-III disease
* Ability to read or understand English
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Subjects, who in the opinion of the principal investigator (PI), may not be able to comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2020-07-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Care coordination | At Baseline
  To test the short and long term effects of the intervention on care coordination (timely appointments and care, use of information to coordinate care, support in managing treatment effects, provides timely information, involvement of family and friends), a 2x2x2 repeated measures analysis of covariance in which the within groups variables are care coordination scores as measured by the Consumer Assessment of Healthcare Providers and Systems Cancer Care Survey at baseline. The between groups measures are the comparisons between 1) study arms, attention control versus intervention, and 2) cancer type, non-small cell lung cancer versus colorectal cancer, with at minimum the baseline care coordination score serving as a covariate. Other covariates may be added to the model pending results of the preliminary analysis.
  Consumer Assessment of Healthcare Providers and Systems Cancer Care Survey, Minimum value = 1 Never ; maximum value = 4 Always, higher is better.
Care coordination | At 4 months
  To test the short and long term effects of the intervention on care coordination (timely appointments and care, use of information to coordinate care, support in managing treatment effects, provides timely information, involvement of family and friends), a 2x2x2 repeated measures analysis of covariance in which the within groups variables are care coordination scores as measured by the Consumer Assessment of Healthcare Providers and Systems Cancer Care Survey at 4 months. The between groups measures are the comparisons between 1) study arms, attention control versus intervention, and 2) cancer type, non-small cell lung cancer versus colorectal cancer, with at minimum the baseline care coordination score serving as a covariate. Other covariates may be added to the model pending results of the preliminary analysis.
  Consumer Assessment of Healthcare Providers and Systems Cancer Care Survey, Minimum value = 1 Never ; maximum value = 4 Always, higher is better.
Care coordination | At 8 months
  To test the short and long term effects of the intervention on care coordination (timely appointments and care, use of information to coordinate care, support in managing treatment effects, provides timely information, involvement of family and friends), a 2x2x2 repeated measures analysis of covariance in which the within groups variables are care coordination scores as measured by the Consumer Assessment of Healthcare Providers and Systems Cancer Care Survey at 8 months. The between groups measures are the comparisons between 1) study arms, attention control versus intervention, and 2) cancer type, non-small cell lung cancer versus colorectal cancer, with at minimum the baseline care coordination score serving as a covariate. Other covariates may be added to the model pending results of the preliminary analysis.
  Consumer Assessment of Healthcare Providers and Systems Cancer Care Survey, Minimum value = 1 Never ; maximum value = 4 Always, higher is better.
Oncologist/primary care providers (PCP) communication | At Baseline
  To test the effect of the intervention on improved communication among oncologists and PCP, a 2x2x2 repeated measures analysis of covariance (AofC) will be used to test for differences on the perceived quality of care coordination and communication by the oncologists and primary care providers (PCPs) treating patients in the attention control arm and intervention arm (between groups), by diagnosis (between groups) at baseline (within group).
  Survey of Physician Attitudes Regarding the Care of Cancer Survivors; minimum value=never; maximum value=always/almost always; higher is better
Oncologist/primary care providers (PCP) communication | At 4 months
  To test the effect of the intervention on improved communication among oncologists and PCP, a 2x2x2 repeated measures analysis of covariance (AofC) will be used to test for differences on the perceived quality of care coordination and communication by the oncologists and primary care providers (PCPs) treating patients in the attention control arm and intervention arm (between groups), by diagnosis (between groups) at 4 months (within group).
  Survey of Physician Attitudes Regarding the Care of Cancer Survivors; minimum value=never; maximum value=always/almost always; higher is better
Oncologist/primary care providers (PCP) communication | At 8 months
  To test the effect of the intervention on improved communication among oncologists and PCP, a 2x2x2 repeated measures analysis of covariance (AofC) will be used to test for differences on the perceived quality of care coordination and communication by the oncologists and primary care providers (PCPs) treating patients in the attention control arm and intervention arm (between groups), by diagnosis (between groups) at 8 months (within group).
  Survey of Physician Attitudes Regarding the Care of Cancer Survivors; minimum value=never; maximum value=always/almost always; higher is better
PCP knowledge in survivorship care | At Baseline
  To test the short and long term effects of the intervention on improved knowledge in survivorship care among primary care providers, a 2x2x2 repeated measures analysis of covariance will be conducted to compare the outcome for the attention control arm and intervention arm (between groups), by diagnosis (between groups) and over time (within groups) with baseline knowledge scores serving as the primary covariate.
  Survey of Physician Attitudes Regarding the Care of Cancer Survivors; minimum value=never; maximum value=always/almost always; higher is better
PCP knowledge in survivorship care | At 4 months
  To test the short and long term effects of the intervention on improved knowledge in survivorship care among primary care providers, a 2x2x2 repeated measures analysis of covariance will be conducted to compare the outcome for the attention control arm and intervention arm (between groups), by diagnosis (between groups) and over time (within groups) with baseline knowledge scores serving as the primary covariate.
  Survey of Physician Attitudes Regarding the Care of Cancer Survivors; minimum value=never; maximum value=always/almost always; higher is better
PCP knowledge in survivorship care | At 8 months
  To test the short and long term effects of the intervention on improved knowledge in survivorship care among primary care providers, a 2x2x2 repeated measures analysis of covariance will be conducted to compare the outcome for the attention control arm and intervention arm (between groups), by diagnosis (between groups) and over time (within groups) with baseline knowledge scores serving as the primary covariate.
  Survey of Physician Attitudes Regarding the Care of Cancer Survivors; minimum value=never; maximum value=always/almost always; higher is better
Survivor outcomes | At Baseline
  Will compare the two arms to determine the efficacy of the intervention on survivor outcomes and analyze using a 2x2x2 repeated measures analysis of covariance. By diagnosis, differences between the attention control and intervention arm participants on responses to the Confidence in Survivorship Information survey measuring patients' knowledge of and self-efficacy in survivorship care will be examined at baseline into the study, controlling for baseline scores on the Confidence in Survivorship Information survey.
  Confidence in cancer Survivorship: minimum value=strongly disagree; maximum value=strongly agree; higher is better
Survivor outcomes | At 4 months
  Will compare the two arms to determine the efficacy of the intervention on survivor outcomes and analyze using a 2x2x2 repeated measures analysis of covariance. By diagnosis, differences between the attention control and intervention arm participants on responses to the Confidence in Survivorship Information survey measuring patients' knowledge of and self-efficacy in survivorship care will be examined at 4 months post enrollment into the study, controlling for baseline scores on the Confidence in Survivorship Information survey.
  Confidence in cancer Survivorship: minimum value=strongly disagree; maximum value=strongly agree; higher is better
Survivor outcomes | At 8 months
  Will compare the two arms to determine the efficacy of the intervention on survivor outcomes and analyze using a 2x2x2 repeated measures analysis of covariance. By diagnosis, differences between the attention control and intervention arm participants on responses to the Confidence in Survivorship Information survey measuring patients' knowledge of and self-efficacy in survivorship care will be examined at 8 months post enrollment into the study, controlling for baseline scores on the Confidence in Survivorship Information survey.
  Confidence in cancer Survivorship: minimum value=strongly disagree; maximum value=strongly agree; higher is better
Patient-centered communication | At Baseline
  To test the short and long term effect of patient-centered communication, a 2x2x2 repeated measure analysis of covariance will be used to test for differences between the attention control arm and intervention arm (between groups), by diagnosis (between groups) using the results from the Patient-Centered Communication survey at baseline , controlling for the baseline measure of patients' perceptions of whether care is centered around their needs.
  Patient-Centered Communication survey; minimum value=never; maximum value=always; higher is better
Patient-centered communication | At 4 months
  To test the short and long term effect of patient-centered communication, a 2x2x2 repeated measure analysis of covariance will be used to test for differences between the attention control arm and intervention arm (between groups), by diagnosis (between groups) using the results from the Patient-Centered Communication survey at 4 months (short-term, primary effect), controlling for the baseline measure of patients' perceptions of whether care is centered around their needs.
  Patient-Centered Communication survey; minimum value=never; maximum value=always; higher is better
Patient-centered communication | At 8 months
  To test the short and long term effect of patient-centered communication, a 2x2x2 repeated measure analysis of covariance will be used to test for differences between the attention control arm and intervention arm (between groups), by diagnosis (between groups) using the results from the Patient-Centered Communication survey at 8 months (long-term, secondary effect) and over time (within groups), controlling for the baseline measure of patients' perceptions of whether care is centered around their needs.
  Patient-Centered Communication survey; minimum value=never; maximum value=always; higher is better
Quality of life: survey | At Baseline
  A 2x2x2 repeated measure analysis of covariance will be used to test for differences by diagnosis between the attention control arm and intervention arm (between groups) using the results from the Functional Assessment of Cancer Therapy - Lung or Functional Assessment of Cancer Therapy - Colorectal Cancer survey at baseline, controlling for the baseline measure of patients' quality of life.
  Functional Assessment of Cancer Therapy - Lung or Functional Assessment of Cancer Therapy - Colorectal Cancer survey Minimum value=0; maximum value=4; higher is better
Quality of life: survey | At 4 months
  A 2x2x2 repeated measure analysis of covariance will be used to test for differences by diagnosis between the attention control arm and intervention arm (between groups) using the results from the Functional Assessment of Cancer Therapy - Lung or Functional Assessment of Cancer Therapy - Colorectal Cancer survey at 4 months (short-term, primary effect) and over time (within groups), controlling for the baseline measure of patients' quality of life.
  Functional Assessment of Cancer Therapy - Lung or Functional Assessment of Cancer Therapy - Colorectal Cancer survey Minimum value=0; maximum value=4; higher is better
Quality of life: survey | At 8 months
  A 2x2x2 repeated measure analysis of covariance will be used to test for differences by diagnosis between the attention control arm and intervention arm (between groups) using the results from the Functional Assessment of Cancer Therapy - Lung or Functional Assessment of Cancer Therapy - Colorectal Cancer survey at 8 months (long-term, secondary effect) and over time (within groups), controlling for the baseline measure of patients' quality of life.
  Functional Assessment of Cancer Therapy - Lung or Functional Assessment of Cancer Therapy - Colorectal Cancer survey Minimum value=0; maximum value=4; higher is better

OTHER OUTCOMES:
Overall reach (participation rate) with primary care providers (Arm I) | Up to 8 months
  Data analysis will be primarily descriptive. Records from the tracking database will be examined and used to understand the extent to which patients' primary care providers assigned to the intervention arm participated in all aspects of the intervention.
Percentage of primary care providers who received a clinical care plan (Arm I) | Up to 8 months
  Data analysis will be primarily descriptive. Data from the tracking database will also be used to understand the percentage of primary care providers who received a clinician care plan.
Primary care providers' use of care plan information for survivorship care (Arm I) | Up to 8 months
  Data analysis will be primarily descriptive. Primary care provider survivor clinical visit notes will also be used to qualitatively assess primary care providers' use of the clinician care plan information to provide quality survivorship care to also understand the level of adoption of the intervention.
Potential barriers and facilitators for intervention implementation and maintenance | Up to 8 months
  Data analysis will be primarily descriptive. Meeting minutes from the quarterly Stakeholder Advisory Council will be qualitatively analyzed to extrapolate data on barriers and facilitators from a clinical, institutional, and implementation (on a systems-level) standpoint.
Outcome Measure for facilitators | Up to 8 months
  Data analysis will be primarily descriptive. Meeting minutes from the quarterly Stakeholder Advisory Council will be qualitatively analyzed to extrapolate data on barriers and facilitators from a clinical, institutional, and implementation (on a systems-level) standpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Sun V, Reb A, Debay M, Fakih M, Ferrell B. Rationale and Design of a Telehealth Self-Management, Shared Care Intervention for Post-treatment Survivors of Lung and Colorectal Cancer. J Cancer Educ. 2021 Apr;36(2):414-420. doi: 10.1007/s13187-021-01958-8. Epub 2021 Jan 8. PMID 33415649

DOCUMENTS (1):
  • Informed Consent Form (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT04428905/ICF_000.pdf